CLINICAL TRIAL: NCT01360294
Title: The Development of a Questionnaire to Assess Symptoms of Small Airways Disease in Patients With Asthma
Brief Title: Development of Small Airway Disease Questionnaire
Acronym: SADQ
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, E. van der Wiel, MD, University Medical Center Groningen
Other Study IDs: SADQ
Record Dates: First submitted 2011-05-12; First posted 2011-05-25 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Asthma
Keywords: Asthma; Small airways disease; Questionnaire
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asthma with small airway disease
- Asthma without small airway disease

SUMMARY:
The aim of this study is to develop a patient reported outcome tool specific to small airways disease, which assesses symptoms and signs of small airways disease and may help in addition to FEF50% to discriminate between asthmatic patients with and without small airways disease.

DETAILED DESCRIPTION:
Inflammation of the small airways contributes to the severity of the disease and affects the quality of life of patients with asthma. However, the exact role and relevance of small airways disease in asthma is still unclear. This is partly due to the difficulty of measuring small airways pathology with a sensitive and specific parameter. The most commonly used variable as an indicator of small airway obstruction is the FEF50%. Currently, it is not known which clinical symptoms are associated with small airways disease and how a patient will perceive small airway abnormalities. This knowledge is important to assess small airways disease in patients with asthma and adjust therapy to improve quality of life.The primary purpose of this study is to develop a questionnaire for patients with asthma with and without small airways disease for general and specialist practice.

ELIGIBILITY:
Inclusion Criteria:

* A doctor diagnosis of asthma
* Age: ≥ 18 and ≤ 75 years
* An FEF50% value that is included in either the lowest or the highest 25th percentile. (Percentiles based on the total asthma patient group present from Asthma/COPD service)

Exclusion Criteria:

* Recent exacerbation of asthma (<2 months) or upper respiration tract infection (<2 weeks)
* Severe airway obstruction at baseline, FEV1pred< 50% or < 1.2L
* Diagnosis of COPD or another pulmonary disease
* Pregnancy or lactating women. (i.e. women of childbearing potential who do not use adequate anticonception as judged by the investigator).
* Restriction, defined as FVC < 80%pred with FEV1/FVC >0.7

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will contain a total of 60 adult patients with asthma, 30 patients with small airways disease and 30 patients without small airways disease.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Symptoms associated with small airways disease | 1 year
  A questionnaire based on symptoms to discriminate between asthmatic patients with and without small airways disease.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands